CLINICAL TRIAL: NCT03229720
Title: Effectiveness of Audio-Visual Distraction Technique Versus Normal Dental Environment for Management of Anxiety in Pediatric Dental Patients, A Randomized Clinical Trial
Brief Title: Evaluation of Audio-Visual Distraction Technique on Child's Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Adel Khalaf Zakhary, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Protocol CairoU
Record Dates: First submitted 2017-07-23; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Anxiety, Dental; Fear, Dental
Keywords: Audio Visual Distraction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician is blinded by naming the groupes into group A and group B
  .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audio-Visual Distraction Group (Active Comparator): In this arm, the patient will be introduced to the audio-visual distraction device and given some instruction on how to use it and rules while using it. other than that, the dental procedure is as same as the other arm group.
  Interventions: Device: Nibiru 3D Virtual Reality Headset
- Normal Dental Environment Group (No Intervention): Normal Dental Environment without any distractions.

INTERVENTIONS:
Device: Nibiru 3D Virtual Reality Headset — This device is a kind of head glass that obstructs the vision with a wide screen showing movies or photos. Earphones are extended from it and inserted in ears. so it obstructs the vision and audio of the surroundings.
  Arms: Audio-Visual Distraction Group

SUMMARY:
Audio-Visual (AV) Distraction is a recent modality introduced to the entertaining market technology for adults and children. Some practitioners started using this modality of distraction in the dental practice to aid in psychological management of patients.

This study is designed to compare between conventional dental visits (No Distraction) and dental visits aided with audio-visual distraction. Providing a safe, comfortable and entertaining dental environment will give pediatric children a better perception regarding the dental environment and motivate them for repetitive dental visits for better dental health care.

DETAILED DESCRIPTION:
[I] Recruitment: Children aged 5~8 years old with teeth decay requiring restorative dental treatment will be randomly selected according to the Intrusion and Extrusion Criteria.

[II] Intervention:

-Steps:

1. The operator will select the teeth; child must have decayed tooth requiring restorative dental treatment.
2. The visit will be started by using the tell-show-do technique to explain the procedure. After that the Facial Image Scale is validated to assess dental anxiety and will be explained to the child. The dentist will ask the child to choose one of the six faces that best represented his/her current emotional state.
3. Pulse oximeter sensor will then be placed and initial pulse rate will be obtained.
4. Patient will choose from a bowl a piece of paper to decide if AV-distraction will be used or not.
5. Above steps will be done in both visits, with and without the intervention.
6. If the toss had AV-distraction, The operator will introduce the Audio-visual device (Virtual Reality Eye Glasses) to the patient and how it works and will allow the patient to choose his favorite show to watch during the dental visit.
7. The operator will instruct the patient with the rules that will be applied during the dental visit to assure complete cooperation.
8. The operator will apply topical and dental anaesthesia
9. Pulse rate will be measured every 5 minutes.
10. The operator will allow extra time if the dental visit ended before the child finishes the tv-show.
11. Then operator will ask the patient to choose from the face scale diagrams about his anxiety state at the end of the visit.

Intervention modifications:

In case the child interrupted the dental visit for questions or any reason, the last record of pulse oximeter will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-8 years old.
* Children with decayed teeth requiring pulp therapy (excluding cases with acute pulpitis)
* Cooperative children and potentially cooperative
* Physically and mentally normal children.
* No previous dental experience involving local anaesthetic administration for the last 2 years

Exclusion Criteria:

* Children with visual impairment.
* Children with hearing disabilities.
* Children with disability complicating the dental treatment as trismus, or TMJ problems.
* Children with highly inflamed pulp tissue inducing pain during dental visit.
* Patients or caregivers who refuse to sign the consent.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Facial Image Scale | Immediately right after the dental visit.
  To measure dental Anxiety by using Facial Image Scale

SECONDARY OUTCOMES:
Oxygen Saturation (using Pulse oximetry) | During the dental visit
  to assess the amount of oxygen saturation and relate to the stress level.

OTHER OUTCOMES:
Heart Rate (using Pulse oximetry) | During the dental visit
  to asses heart beats per minute and relate it to the patient's anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hamdy, Professor, Study Director — Cairo University; Nada Wassef, Ass. Prof, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided